CLINICAL TRIAL: NCT05490225
Title: A Study to Evaluate the Safety and Effectiveness of Voyager's Access Device for Patients Undergoing Routine Hemodialysis (Access Cannulation Trial II)
Brief Title: Access Cannulation Trial II
Acronym: ACT II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Voyager Biomedical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Access Cannulation Trial II
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Dialysis; Complications; Vascular Access Complication

STUDY DESIGN:
Intervention Model Description: This is a pivotal, interventional, prospective, single arm, open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Ark Implantation (Experimental): Single arm study. Depending on the clinical needs of the patient, the physician will decide if a single return device is needed (ex. easily cannulatable arterial pull site but the venous return access site is poorly accessible for cannulation) or two devices (both arterial pull and venous return are poorly accessible for cannulation).
  Interventions: Device: VenaSure

INTERVENTIONS:
Device: VenaSure — The device will be surgically implanted at the access site in subjects undergoing routine hemodialysis. The device is expected to provide a target to aid in long-term cannulation success.

SUMMARY:
This is a pivotal, interventional, prospective, single-arm, open-label, multi-site clinical investigation intended to support FDA clearance of the study device based on the safety and efficacy of the device in cannulating arteriovenous fistulas (AVFs) for hemodialysis procedures.

DETAILED DESCRIPTION:
This clinical investigation is estimated to last approximately 48-60 months, from initial participant enrollment until all data collection is complete on the final participant. After the patient has the study device implanted, they will be observed for 6 weeks as the implant site heals. The patient will be monitored for 36 months after device implantation as they undergo routine dialysis. Subjects will exit the investigation after the last visit and no device-related adverse events have been identified or are being monitored

ELIGIBILITY:
Inclusion:

1. The subject's AVF is deemed uncannulatable because:

   1. The subject's anticipated cannulation zone(s) is/are >6mm in depth from the surface of the skin to the anterior wall of the access vein as confirmed by ultrasound within 8 weeks prior to device implantation (each zone, Arterial/Pull and Venous/Push, shall be assessed independently of one another for device placement):

      * Arterial/Pull Zone: _____ mm deep
      * Venous/Push Zone: _____ mm deep

      OR
   2. The subject's dialysis unit (which includes an experienced cannulator) attests that repeated cannulation is not achievable in their clinic due to one of the following:

      * Failed access attempt in a fistula that was previously approved for cannulation, or
      * Unable to palpate the fistula such that cannulation is not possible without patient risk.
2. The access surgeon caring for the subject attests that the device is likely to be at least equivalent to other methods (such as venous transposition or suction-assisted lipectomy) that could make the AVF easier to access and reduce risk of cannulation infiltrations.
3. The subject has either a radio-cephalic, brachio-cephalic or transposed brachio-basilic fistula.

Exclusion:

1. The subject's access vein is >15mm in depth at either cannulation zones as measured by ultrasound within 8 weeks prior to device implantation.

   * Arterial/Pull Zone: _____ mm in depth
   * Venous/Push Zone: _____ mm in depth Note: these values should match inclusion criteria #1
2. Both bidimensional measurements in the subject's access vein have a diameter of <4mm, taken with a tourniquet in place or through manual compression to the outflow, as measured by ultrasound within 8 weeks prior to device implantation (cannulation zone specific - one zone does not affect the other's eligibility).

   * Arterial/Pull Zone: _____ x _____ mm in diameter
   * Venous/Push Zone: _____ x _____ mm in diameter
3. The subject has a flow rate of <550mL/min in the inflow artery proximal to the arterial anastomosis as measured by ultrasound within 8 weeks prior to device implantation.

   • Flow: _____ mL/min
4. The subject does NOT have a prescription to receive maintenance hemodialysis at least 2 times per week.
5. The subject's life expectancy is <1 year per the Investigator.
6. The subject does NOT have a signed and dated consent form.
7. The AVF is a non-transposed basilic or brachial vein outflow AVF.
8. The subject has high flow rates placing them at risk for heart failure and death at the discretion of the Investigator.
9. The subject has a known skin infection, hypersensitive skin, skin breakdown/erosion or skin allergies at the potential implant sites.
10. The subject has a known active systemic infection or positive blood cultures present.
11. The subject's AVF has undergone a major revision and at the discretion of the Investigator can impact fistula viability and device placement (such as DRIL or PTFE segment insertion, banding, aneurysm repair, etc.), or the subject has had an occurrence of and/or intervention for AV access stenosis or thrombosis within the past month (excluded to avoid unnecessary placement into an AVF with a high likelihood of failure).
12. The subject is <18 years of age.
13. The subject plans to become pregnant prior to their potential treatment date.
14. The subject has a body mass index >50kg/m2.
15. The subject has a known clinically significant bleeding or coagulation disorder, including but not limited to low platelet count (<50,000), hypercoagulable state (e.g., antithrombin IE deficiency, antiphospholipid or anticardiolipin antibodies, Factor V Leiden, circulating Lupus anticoagulant, current, heparin-induced thrombocytopenia, protein C or S deficiency, history of recurrent deep vein thrombosis not related to AV access).
16. The subject has an active malignancy.
17. The subject has a known or suspected allergy to titanium, aluminum, or vanadium.
18. The subject has had a significant cardiovascular event/intervention that makes them a poor surgical candidate such as myocardial infarction, angioplasty, or stent placement within 3 months of implantation.
19. The subject has had a significant peripheral vascular disease requiring a major intervention within the previous 12 months (in the target limb).
20. The subject has had a significant neurovascular event such as stroke or major intervention within the previous 12 months.
21. The subject has an uncontrolled major symptomatic medical problem per the Investigator.
22. The subject has a likelihood of poor protocol compliance due to mental incapacity, an inability to understand treatment instructions, or for any other reason in the opinion of the Investigator.
23. The subject is currently participating in another investigational drug or device investigation that could clinically interfere with the endpoints of this investigation.
24. The subject's conversion to home hemodialysis is anticipated at any point during their foreseeable participation in this investigation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-23 (Actual); Primary Completion 2027-03-25 (Estimated); Study Completion 2027-03-25 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the effectiveness of the study device in facilitating cannulation of arteriovenous fistulas (AVFs) for hemodialysis. | 6 months
  Incidence of success for achieving clinically functional access within a 6-month timeframe from approved cannulation through the study device.
To evaluate the safety of the study device. | 12 months
  The assessment and occurrence of device-related, serious adverse events (SAEs) of clinical interest (infection, aneurysm, complicated seroma) during a 12- month follow-up period from initial implantation adjudicated by a Data Monitoring Committee (DMC)

SECONDARY OUTCOMES:
To investigate time-related parameters surrounding the study device in facilitating hemodialysis. | 12 months
  Cumulative duration (days) of hemodialysis catheter exposure (post device implantation), including CVC reinsertion events
To further evaluate the safety of the study device | 12 months
  Incidence and types of device-related complications
To further evaluate the safety of the study device | 12 months
  Days to successful cannulation and hemodialysis through the device
To further evaluate the safety of the study device | 6mo from approved cannulation through the device
  Vascular access interventions required to achieve the primary effectiveness endpoint
To further evaluate the safety of the study device | 36 months
  Time required to achieve the primary endpoint for all evaluable subjects.
To further evaluate the safety of the study device | 3 months, 6 months, 12 months
  (Post intervention) Functional Cumulative Patency utilizing Kaplan-Meier methodology
To further evaluate the safety of the study device | 4 weeks from initial implantation
  Initial Safety Assessment (Time Frame = 4 weeks from initial implantation) adjudicated by a Data Monitoring Committee (DMC).

OTHER OUTCOMES:
Exploratory Outcome 1 | 36 months
  Infiltration rate and AVF failure rate after infiltration
Exploratory Outcome 2 | SCRN/BSLN, 6 months, 12 months
  Patient Satisfaction Survey
Exploratory Outcome 3 | 12 months
  Utilization of health care resources: health economic data analysis to be performed based on available study data for the treatment related costs (e.g. procedural costs, hospital costs, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Hohmann, MD, Principal Investigator — Baylor Scott and White Health
Locations (8):
- United States (8):
  - Trinity Research Group, Dothan, Alabama
  - Apex Research, Riverside, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Northwell Health, Hyde Park, New York
  - MUSC Health Orangeburg, Orangeburg, South Carolina
  - Cardiothoracic and Vascular Surgeons, Austin, Texas
  - Baylor Scott & White, Dallas, Texas
  - Fairlawn Surgery Center, Roanoke, Virginia

IPD SHARING:
Plan to Share IPD: No
If data is shared after study completion it will be redacted of any PHI

REFERENCES:
- See also: Related Info — http://www.voyagerbiomedical.com